CLINICAL TRIAL: NCT05397262
Title: Register-Trial Based on an Agreement of Health Insurances With the Department of Radiation Therapy of the University Hospital Erlangen for the Application of Regional Hyperthermia in Bladder Cancer: Organ-preservative Therapy of Bladder Cancer With Radiotherapy or Radiochemotherapy Combined With Hyperthermia
Brief Title: Organ-preservative Therapy of Bladder Cancer With Radiotherapy or Radiochemotherapy Combined With Hyperthermia
Acronym: HyBla_RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Oliver J. Ott, Principle Investigator, University of Erlangen-Nürnberg Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HyBla_RCT
Record Dates: First submitted 2017-04-10; First posted 2022-05-31 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; Hyperthermia; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Hyperthermia | interventions — Diathermy; Hyperthermia, Induced; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard Arm (Other): 1 Arm: combination Treatment: Deep regional hyperthermia: 1-2/week up to 10 sessions Radiotherapy: 50.4Gy + Boost 5.4Gy (R0) or 9.0Gy (R1/2)
  Chemotherapy:
  5-Fluorouracil 600mg/m^2, civ 120h; d1-5, 29-3
  Chemotherapy:
  Cisplatin 20mg/m^2; d1-5, 29-33
  Interventions: Other: Hyperthermia; Radiation: Radiotherapy; Drug: Chemotherapy 5-Fluorouracil; Drug: Chemotherapy Cisplatin

INTERVENTIONS:
Other: Hyperthermia — Deep Regional Hyperthermia (RHT) 1-2/week up to 10 sessions a type of cancer treatment in which body tissue is exposed to high temperatures (up to 113°F).
  Other Names: Thermal therapy or thermotherapy
Radiation: Radiotherapy — 50,4 Gy (28 x 1,8 Gy) plus Boost: If R0: 5,4 Gy; If R1/2: 9 Gy
Drug: Chemotherapy 5-Fluorouracil — 600 mg/m^2 civ 120h; d 1-5, 29-33
Drug: Chemotherapy Cisplatin — 20 mg/m^2; d1-5, 29-33

SUMMARY:
Analysis of the efficacy and the compatibility of deep regional hyperthermia in combination with radiotherapy and chemoradiotherapy in bladder cancer

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed bladder cancer
* M0
* ECOG-performance status ≤ 2
* Informed consent

Exclusion Criteria:

* Pre-existing uncontrolled cardiac disease, signs of cardiac failure, or rhythm disturbances requiring therapy
* Cardiac Pacemaker
* Myocardial infarction within the past 12 months
* Congestive heart failure
* Complete bundle branch block
* New York Heart Association (NYHA) class III or IV heart disease
* Disease that would preclude TUR, chemoradiation or deep regional hyperthermia
* Metal implants (lenght > 2cm or dense clusters of marker clips in the pelvis)
* Active or therapy-resistent bladder infections
* Pre-existing or concommitant immunodeficiency Syndrom
* Pregnant or lactating women
* Patients not willing to use effective contraception during and up to 6 months after therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-03-29 (Actual); Primary Completion 2098-12-31 (Estimated); Study Completion 2099-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Participants will be followed for up to 5 years after the end of therapy
  Overall survival

SECONDARY OUTCOMES:
Bladder preservation rate | Participants will be followed for up to 5 years after the end of therapy
  Rate of patients where bladder can be preserved
Disease free survival | Participants will be followed for up to 5 years after the end of therapy
  Length of survival without disease recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Ott, MD, Principal Investigator — Dept. of Radiation Therapy, University Hospital Erlangen
Locations (1):
- Dept. of Radiation Therapy, University Hospital Erlangen, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Undecided